CLINICAL TRIAL: NCT01522560
Title: Evaluation of Multiscore Feedback in Professionalism for Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11-473
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2017-08

CONDITIONS: CA2 and CA3 Residents Doing a Two Month Rotation in; Pediatric Anesthesia Department
Keywords: CA2 and CA3 residents; Pediatric Anesthesia
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Residents will be randomly assigned to a feedback group or to the control group. Besides the standard evaluation at the end of the rotation, in both groups, residents will receive every week a MSF evaluation from the faculty, the patients' parent, and the coworker. Also, for every resident a baseline self assessment will be applied at the beginning and at the end of the rotation. Only the group assigned to feedback is going to have a 'coaching meeting' every month with the Chairman of Department of Pediatric Anesthesia to identify strengths and weaknesses and create strategies for improvement, based on the MSF.
  Interventions: Other: Control group
- Feedback group (Active Comparator): Residents will be randomly assigned to a feedback group or to the control group. Besides the standard evaluation at the end of the rotation, in both groups, residents will receive every week a MSF evaluation from the faculty, the patients' parent, and the coworker. Also, for every resident a baseline self assessment will be applied at the beginning and at the end of the rotation. Only the group assigned to feedback is going to have a 'coaching meeting' every month with the Chairman of Department of Pediatric Anesthesia to identify strengths and weaknesses and create strategies for improvement, based on the MSF.
  Interventions: Other: Feedback group

INTERVENTIONS:
Other: Feedback group — Besides the standard evaluation at the end of the rotation, in both groups, residents will receive every week a Multiscore Feedback (MSF) evaluation from the faculty, the patients' parent, and the coworker. Also, for every resident a baseline self assessment will be applied at the beginning and at the end of the rotation.
  This group is going to have a 'coaching meeting' every month with the Chairman of Department of Pediatric Anesthesia to identify strengths and weaknesses and create strategies for improvement, based on the Multiscore Feedback (MSF).
  Arms: Feedback group
Other: Control group — Besides the standard evaluation at the end of the rotation, in both groups, residents will receive every week a Multiscore Feedback (MSF) evaluation from the faculty, the patients' parent, and the coworker. Also, for every resident a baseline self assessment will be applied at the beginning and at the end of the rotation.
  Arms: Control Group

SUMMARY:
Professionalism is one of the six competences required by The Accreditation for Graduate Medical Education Outcome Project to be taught and evaluated during residency. Anesthesia residents are faced with unique communication challenges in their practice including brief contact time with their patients, operating room efficiency pressure, etc. To assess professionalism in Anesthesiology residents is important to obtain evaluations from people with whom they interact including patients, surgeons, colleagues and members of the support team. The Multisource feedback (MSF) approach has been used to evaluate communication skills and professionalism among practicing physicians and residents in a variety of settings. This evaluation model has never been used previously to evaluate anesthesia residents. The investigators propose a randomized controlled trial to validate and evaluate a MSF in professionalism for anesthesia residents. Participants include eighty residents doing two months rotation in Pediatric Anesthesia Department at The Cleveland Clinic Anesthesia Institute from July 1, 2011 and June 30, 2013. MSF questionnaires will be validated using face and content validity methods and comparing them with the current system of evaluation. Residents will be randomly assigned to a feedback group or to the control group. Both groups will receive MSF evaluation from the faculty, patients' parent and coworker. Only the group assigned to feedback is going to have a 'coaching meeting' every month to identify strengths and weaknesses and create strategies for improvement. The investigators are planning to compare the mean values of the baseline evaluations with the mean values obtained after the first and second months from the MSF.

ELIGIBILITY:
Inclusion Criteria:

* CA2 and CA3 residents doing a two month rotation in Pediatric Anesthesia Department

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Validate Multiscore Feedback (MSF) | up to 60 days
  To evaluate content validity, copies of the questionnaires will be sent to experts in education in the Anesthesia Institute and Graduate Medical Education at The Cleveland Clinic; they will be asked if the new questionnaires are a good tool to measure professionalism for anesthesia residents

SECONDARY OUTCOMES:
secondary goal is to test a Multiscore Feedback (MSF) as a method of evaluation in professionalism for anesthesia residents. | up to 18 months
  We will assess the impact of feedback using the MSF (versus no feedback) on the professional behavior of anesthesia residents as measured by the MSF. The randomized groups of residents with and without feedback will be compared on mean MSF score after the first and second months of the rotation using a linear mixed effects model to account for the correlation between measurements on the same resident and to adjust for baseline score as a covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Riveros, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States